CLINICAL TRIAL: NCT01620281
Title: The no!no!Back Continuous Passive Motion Device for the Treatment of Chronic Low Back Pain: A Randomized Controlled Pilot Study
Brief Title: The Efficacy of the no!no!Back for Chronic Low Back Pain
Acronym: LBP-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radiancy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBP-1
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Mild to Moderate Chronic Low Back Pain
Keywords: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate treatment (IT) (Experimental): Subjects from this group will receive the device immediately. Subjects will be instructed to treat themselves daily for 3 weeks, in up to three 10-minutes sessions. All subjects will receive a diary to record details of the daily use of the device (time of day, position of legs, and number of daily uses), degree of pain, a weekly ODI questionnaire, and record of any back/pain related events. After 3 weeks the subjects from the IT group will return the device and at 6 weeks they will visit again for the final evaluation.
  Interventions: Device: no!no!Back
- Waiting List Control (WLC) (Other): The WLC group will go through the same evaluations at the same time intervals but will begin treatments 3 weeks later during which they will fill the diary daily but not use the device.
  Interventions: Device: no!no!Back

INTERVENTIONS:
Device: no!no!Back — Self treatments daily for 3 weeks, in up to three 10-minutes sessions

SUMMARY:
This pilot study is designed to evaluate the efficacy of the no!no!Back continuous passive motion device in relieving of mild to moderate non-specific low back pain.

DETAILED DESCRIPTION:
The no!no!Back is an electrically operated, continuous passive motion device including a platform that performs angular oscillations. The device is intended to be used at home as an accessory for relieving of mild to moderate low back pain (LBP).

This study is designed to determine the efficacy of daily use home use with the no!no!Back device during 3 weeks and to assess the sustained effect 3 weeks later. Up to 30 subjects will be randomized to either an immediate treatment (IT) group that will receive the no!no!Back device at the baseline visit, or to the wait-list control (WLC) group that will receive the device 3 weeks later. The evaluation will include level of pain using the numerical rating scale (NRS), functional health status by Oswestry disability index (ODI), and subject satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 or more
* Level of pain - mild to moderate low back pain (≤5 NRS pain)
* Chronic - symptoms must have been present for at least 12 weeks or more.
* Location - lower tip of scapula to back of pelvis
* Etiology - non-specific

Exclusion Criteria:

* Patients who have low back pain due to specific and known etiological causes (infection, tumor, osteoporosis, ankylosing spondylitis, fracture, inflammatory process, radicular syndrome, cauda equinal syndrome).
* Pregnant or lactating
* Recent history of violent trauma
* History of previous back surgery
* Constant progressive, non mechanical pain (no relief with bed rest)
* Chronic pain other than low back pain
* Past medical history of malignant tumour
* Has taken an investigational drug within the past 30 days prior to entering the study, or currently enrolled in another investigational study
* Mental disorder that would lead to difficulty in questionnaire completion
* Current or future litigation for low back pain
* Prolonged use of corticosteroids
* Physical disability that prevents the subject to lie down/get up
* Drug abuse, immunosuppression, HIV
* Any other condition which in the physician's opinion would make it unsafe for the subject to be treated.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in pain level after 3 weeks compared to baseline (before treatment) | 3 weeks
  Pain level will be scored by the subject using a numerical rating scone on a 0 to 10 scale where 10 represents the highest degree of pain and 0 represents a complete lack of pain

SECONDARY OUTCOMES:
Change in functional health status by ODI | 3,6 weeks
  Functional health status will be determined by the ODI questionnaire filled by the subject (10 multi-choice questions, takes 5 minutes to answer).
Subject satisfaction | 6 weeks
  The subject will be verbally asked to grade his/her overall satisfaction according to the satisfaction assessment scale based on a 5-point Likert scale detailed in Table 3 where 0 represents very unsatisfied and 4 represents very satisfied. In addition the subject will fill a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lilach Gavish, PhD, Study Director — Friedman Skin & Laser Center; David J Friedman, MD, Principal Investigator — Friedman Skin & Laser Center
Locations (1):
- Koren Physiotherapy Institute, Mevaseret Zion, Israel

REFERENCES:
- [Derived] Gavish L, Barzilay Y, Koren C, Stern A, Weinrauch L, Friedman DJ. Novel continuous passive motion device for self-treatment of chronic lower back pain: a randomised controlled study. Physiotherapy. 2015 Mar;101(1):75-81. doi: 10.1016/j.physio.2014.06.003. Epub 2014 Jul 28. PMID 25280603